CLINICAL TRIAL: NCT01273285
Title: Reproducibility of Nerve Fiber Layer Thickness Measurements in Patients With Glaucoma and Healthy Controls Using Spectral-Domain and Time-Domain OCT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Funk Jens, Prof. Dr. Dr., University hospital Zurich, AUG Augenklinik
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RNFL-Repro
Record Dates: First submitted 2011-01-07; First posted 2011-01-10 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Glaucoma Patients and Healthy Controls
MeSH Terms: interventions — Proton Therapy

INTERVENTIONS:
Device: Spectralis® SD-OCT, Heidelberg Engineering GmbH, H

SUMMARY:
To assess the reproducibility of Spectral-Domain-OCT (SD-OCT) retinal nerve fiber layer thickness (RNFL) thickness measurements in healthy volunteers and patients with glaucoma and to compare these results to conventional Time-Domain-OCT (TD-OCT).

* Trial with medical device

ELIGIBILITY:
Inclusion criteria: control group:

age 18yo or older, healthy

glaucom group: age 18yo or older, diagnosis of primary open angle glaucoma (POAG)

Exclusion criteria: Exclusion criteria in the control group were history of glaucoma, history of any other ocular disease, or intraocular pressure greater than 21mmHg. Exclusion criteria in the glaucoma group were history of other optic neuropathies.

or severe optic media opacities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
reproducibility of retinal nerve fiber layer thickness measurement

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- Zurich, Switzerland

REFERENCES:
- [Derived] Toteberg-Harms M, Sturm V, Knecht PB, Funk J, Menke MN. Repeatability of nerve fiber layer thickness measurements in patients with glaucoma and without glaucoma using spectral-domain and time-domain OCT. Graefes Arch Clin Exp Ophthalmol. 2012 Feb;250(2):279-87. doi: 10.1007/s00417-011-1811-9. Epub 2011 Sep 10. PMID 21909812